CLINICAL TRIAL: NCT06670664
Title: Head Start REACH: Strengthening Outreach, Recruitment, and Engagement Approaches with Families
Acronym: HeadStartREACH
Status: Not yet recruiting | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Brazelton Touchpoints Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: HeadStartREACH2
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-07

CONDITIONS: Head Start Recruitment, Selection, and Enrollment Practices

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Head Start Program: Recruited Head Start program and its program director, a staff member in charge of recruitment, selection, and enrollment, and community partners who help support those efforts, and parents/caregivers of students enrolled in one classroom.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. This is a single-group study.

SUMMARY:
Mathematica, funded by the Administration for Children and Families (ACF) Office of Planning, Research, and Evaluation (OPRE) in the U.S. Department of Health and Human Services (HHS) will conduct a one-time mixed-methods study to improve understanding about Head Start programs' practices for recruitment, selection, and enrollment of families experiencing adversities. Using data gathered from surveys and focus groups, this study aims to provide in-depth contextual information about recruitment, selection, and enrollment practices and experiences; identify promising practices; and inform training and technical assistance (T/TA) regarding recruitment, selection, and enrollment challenges and needs.

Data collection will occur in fall 2024. The study team will field surveys with Head Start staff from up to 60 Head Start programs; parents/caregivers from those 60 programs, and staff from up to 180 community partner organizations that work with those 60 Head Start programs. We will also conduct focus groups with the eligibility, recruitment, selection, enrollment, and attendance (ERSEA) lead staff from some of the programs.

DETAILED DESCRIPTION:
The purpose of this mixed-methods study is to expand understanding of how Head Start programs implement, recruitment, selection, and enrollment practices and how such practices reflect their community contexts. Using survey data collected from Head Start staff, enrolled families, and community partner organizations, the study aims to provide in-depth contextual information about Head Start programs' recruitment, selection, and enrollment practices and experiences; identify promising practices; and inform T/TA regarding recruitment, selection, and enrollment challenges and needs. Ultimately, this study seeks to share information with the wider field about promising practices to improve the recruitment, selection, and enrollment of families, including those experiencing adversities. The study will supplement the survey data with qualitative data collected through focus groups with Head Start ERSEA lead staff.

The investigators propose the following data collection activities, to be carried out in fall 2024:

1. A program director web survey: To obtain information about staff to guide the selection of ERSEA lead staff and community partners for the ERSEA lead staff survey and community partner organization staff survey. To obtain information about the characteristics of the families in the program and community, and program's enrollment numbers.
2. An ERSEA lead staff web survey: To obtain information to understand a program's use, perceived effectiveness of, and challenges with recruitment, selection, and enrollment practices; identify promising practices for replication.
3. A community partner web survey: To obtain information to understand how community partner organization staff support the recruitment, selection, and enrollment of families into Head Start programs.
4. A parent/caregiver survey that can be completed on paper or via the web: Obtain information about characteristics of families enrolled in Head Start and understand their reasons for choosing Head Start, as well as their experiences with and perceptions of recruitment, selection, and enrollment practices.
5. A semi-structured focus group guide for ERSEA lead staff: Obtain information to understand the perceived effectiveness of recruitment, selection, and enrollment practices; understand promising practices for replication.

ELIGIBILITY:
Inclusion Criteria:

* Program director at Head Start program
* ERSEA staff members at Head Start program
* Staff at community partner organizations that work with Head Start program
* Families enrolled in Head Start program

Exclusion Criteria:

* Does not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Head Start program directors; Head Start staff involved in implementing recruitment, selection, and enrollment activities; staff in community organizations with which the Head Start program partners to serve families eligible for Head Start; families who are enrolled in Head Start programs.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-09-24 (Estimated)

PRIMARY OUTCOMES:
Head Start Program Directors Survey - Program characteristics of the purposive sample | 1 month
  Study-developed survey instrument will collect data on Head Start program characteristics and the characteristics of the families the program serves. Will also collect roles and contact information for ERSEA lead staff members and staff members from community partner organizations so these respondents can be invited to complete their respective surveys. Conduct descriptive analysis of survey data to report program and community characteristics.
ERSEA Lead Staff Survey on Recruitment, Selection, and Enrollment Practices of purposive sample of programs | 1 month
  Study-developed survey instrument will collect data on respondent and Head Start program background characteristics; staffing and staff training related to recruitment, selection, and enrollment; development and use of recruitment, selection, and enrollment practices. Study will use the data to measure and report on program recruitment, selection, and enrollment practices in the community.
Community Partner Organization Staff Survey on Partnerships with purposive sample of Head Start programs | 1 month
  Study-developed survey instrument will collect data on the community partner organization characteristics; its partnership and communication with Head Start; and activities and training for connecting eligible families to Head Start. Study will use the data to measure and report on how community partners support Head Start recruitment, selection, and enrollment practices.
Head Start Parent/Caregiver Survey on Head Start Recruitment and Enrollment Experiences with purposive sample of Head Start programs | 1 month
  Study-developed survey instrument will collect data on family background and demographics as well as family experience with recruitment into Head Start; their experience with the waitlist; their experience enrolling into Head Start; and their overall experience with Head Start program supports and services. Study will use the data to measure and report on families' experiences with program recruitment, selection, and enrollment practices.
Focus Group Guide for Convenience Sample of ERSEA Lead Staff on Recruitment, Selection, and Enrollment Practices from purposive sample of Head Start programs | 1 month
  Study-developed qualitative protocol will collect data on ERSEA lead staff experience with developing and using recruitment, selection, and enrollment practices and which practices they found to be successful with families experiencing adversities. Study will use the data to measure and report on contextual information related to program recruitment, selection, and enrollment practices in the community.

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Tarullo, EdD, Principal Investigator — Mathematica Policy Research, Inc.

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the study's four surveys will be transmitted to the Child & Family Data Archive or a similar data archive as restricted use data files at the end of the study so it can be used by other researchers. The de-identified datasets will only include data related to study objectives and outcomes.
Supporting Information: Study Protocol, ICF
Time Frame: Starting approximately four months after study publication is complete.
Access Criteria: Access to the de-identified datasets will be controlled and overseen by the Child and Family Data Archive (or similar data archive). The datasets from this study will be restricted use data, which require an application process to access.

REFERENCES:
- [Background] Baxter, C, N. Aikens, L. Tarullo, C. Ayoub, J. Roberts, C. Mondi-Rago, and M. I. Gaither. "Recruitment, Selection, Enrollment, and Retention Strategies with Head Start-Eligible Families Experiencing Adversity: A Review of the Literature." OPRE Report #2022-97. Washington, DC: Office of Planning, Research, and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services, 2022.
- [Background] Shah, H, T. Shenbanjo, C. Lauver, K. St. Kitts, N. Aikens, and L. Tarullo. "Strengthening Outreach, Recruitment, and Engagement Approaches with Families: The Head Start REACH Case Study Report." OPRE Report #2023-132. Washington, DC: Office of Planning, Research, and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services, 2023.
- [Background] Shah, H., and L. Tarullo. "Reaching and Supporting Families Most in Need: Lessons and Practice Considerations from the Head Start REACH Case Studies." OPRE Report #2023-295. Washington, DC: Office of Planning, Research, and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services, 2023.